CLINICAL TRIAL: NCT04388176
Title: A Phase 2, Single-center, Randomised, Double-blind, Placebo-controlled, Cross-over Cold Challenge Study Investigating the Effect of C21 on Cold-induced Vasoconstriction in Subjects With Raynaud's Phenomenon (RP) Secondary to Systemic Sclerosis (SSc)
Brief Title: Cold Challenge With C21 in RP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VP-C21-004; 2019-003203-35 (EudraCT Number)
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-07

CONDITIONS: Raynaud Phenomenon; Systemic Sclerosis
Keywords: Systemic sclerosis; Raynaud's phenomenon; Vasoconstriction
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic | interventions — compound 21

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, placebo-controlled cold challenge study. A cross-over design is applied to control for inter-individual variability in response to cold challenge.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be conducted in double-blind fashion and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C21 followed by placebo (Experimental)
  Interventions: Drug: C21; Drug: Placebo
- Placebo followed by C21 (Experimental)
  Interventions: Drug: C21; Drug: Placebo

INTERVENTIONS:
Drug: C21 — C21 as first treatment
  Arms: C21 followed by placebo
Drug: C21 — C21 as second treatment
  Arms: Placebo followed by C21
Drug: Placebo — Placebo as second treatment
  Arms: C21 followed by placebo
Drug: Placebo — Placebo as first treatment
  Arms: Placebo followed by C21

SUMMARY:
This is a randomised, double-blind, placebo-controlled, cross-over phase 2 trial investigating the effect of C21 on cold-induced vasoconstriction in subjects with Raynaud's phenomenon secondary to systemic sclerosis. The purpose of the trial is to achieve a vasodilatory effect in subjects with Raynaud's phenomenon by stimulation of the AT2R (angiotensin II type 2 receptor) with C21.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any trial related procedures are performed.
2. Subjects diagnosed with SSc according to European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria
3. Age 19-75 years inclusive
4. RP secondary to SSc as determined by the investigator, and with a typical frequency of attacks during the winter months (November-March) of on average at least 5 per week.

Exclusion Criteria:

1. Smoking (including E-cigarettes) or use of nicotine replacement therapy for three months prior to Visit 1 and during the trial.
2. BMI >30
3. Mixed connective tissue disease or "overlap" (i.e. those who satisfy more than one set of ACR criteria for a rheumatic disease).
4. Concurrent serious medical condition with special attention to cardiac or ophthalmic conditions which in the opinion of the investigator makes the patient inappropriate for this study
5. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma and cervical intraepithelial neoplasia grade I
6. Planned major surgery within the duration of the study
7. Subjects who forsake any alcohol intake or have known uncontrolled allergic conditions or allergy/hypersensitivity to any components of the trial drug or placebo excipients (see Section 7.1)
8. Blood donation (or corresponding blood loss) within three months prior to Visit 1
9. Treatment with any of the medications listed below within 4 weeks prior to Visit 1:

   * Any dose-change or initiation of vasoactive substances

     , and not able or willing to withhold these medications for 3 days preceding Visit 2 and Visit 3, respectively
   * Iloprost
   * Any treatment with CYP3A4 inducers (e.g. rifampicin, phenytoin, St John's Wort)
   * Any treatment with CYP3A4 inhibitors (e.g. clarithromycin, ketoconazole, nefazodone, itraconazole, ritonavir)
   * Any treatment with medicines that are substrates of CYP1A2, CYP3A4 or CYP2C9 with a narrow therapeutic range
   * Any experimental drug
   * Any systemic immunosuppressive therapy other than:

     * Inhaled corticosteroids which can be used throughout the trial period
     * The continuation of stable doses of <10 mg prednisolone
     * Mycophenolate mofetil (MMF) which must be withheld for 3 days preceding Visit 2 and Visit 3
10. Any of the following findings at the time of screening:

    * Finger temperature below 27°C after acclimatising at an ambient temperature of 23°C for a period of 20 minutes
    * Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG, as judged by the Investigator
    * Positive results for HBsAg, HCVAb or HIV 1+2 Ag/Ab
    * Positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG)
    * Clinically significant abnormal laboratory value at Visit 1 indicating a potential risk for the subject if enrolled in the trial as evaluated by the Investigator
11. Pregnant or breast-feeding female subjects.
12. Female subjects of childbearing potential not willing to use contraceptive methods described in Section 5.3.1.
13. Male subjects not willing to use contraceptive methods described in Section 5.3.1.
14. Participation in any other interventional trial during the trial period
15. Subjects known or suspected of not being able to comply with this trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Herrick, MD, Principal Investigator — Department of Rheumatology Salford Royal Hospital, Manchester,United Kingdom
Locations (1):
- Department of Rheumatology, Salford Royal Hospital, Manchester, Salford, United Kingdom

REFERENCES:
- [Derived] Herrick AL, Batta R, Overbeck K, Raud J, Manning J, Murray A, Dinsdale G, Tornling G. A phase 2 trial investigating the effects of the angiotensin II type 2 receptor agonist C21 in systemic sclerosis-related Raynaud's. Rheumatology (Oxford). 2023 Feb 1;62(2):824-828. doi: 10.1093/rheumatology/keac426. PMID 35894657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial planned to include 16 subjects, however as recruitment was challenging during the COVID-19 (coronavirus disease 2019) pandemic, enrolment was stopped prematurely when 12 subjects were randomised. This ensured that trial results could be available in a timely manner.
Pre-assignment Details: A total of 20 unique subjects provided informed consent and were enrolled in the trial. Seven of these were screening failures. In addition, 2 subjects were not randomised; 1 subject due to the COVID-19 pandemic and 1 subject due technical issues with the Holter ECG. The latter subject was re-screened. A total of 12 subjects were randomised.
Period: Overall Study
Arm/Group | C21 Followed by Placebo | Placebo Followed by C21
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C21 Followed by Placebo | Placebo Followed by C21 | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [46 to 69] | 51.5 [35 to 67] | 55.5 [35 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 12
Height [Mean (Full Range); unit: cm] | 163.1 [154.0 to 180.0] | 164.3 [155.0 to 171.5] | 163.7 [154.0 to 180.0]
Weight [Mean (Full Range); unit: kg] | 68.3 [50.8 to 90.0] | 64.9 [54.0 to 79.8] | 66.6 [50.8 to 90.0]
BMI [Mean (Full Range); unit: kg/m^2] | 25.6 [20.2 to 29.0] | 24.2 [19.2 to 29.3] | 24.9 [19.2 to 29.3]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Rewarming of Each Finger After Cold Challenge (AUC) as Measured by Thermography
Description: Area under the curve for rewarming of each finger after cold challenge as measured by thermography for 15 min
Time Frame: For 15 min after cold challenge (40-55 min after IMP [investigational manufacturing product] administration)
Population: Full analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: C*sec
Groups:
- Placebo: A single oral dose of placebo
- C21 200 mg: A single oral dose of 200 mg C21
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
C*sec | 19558.43 (4.36) | 20045.96 (7.68)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Test type: Equivalence — Differences in treatment groups in the primary endpoint (log (AUC)) was to be detected with a power of 90% and alpha=0.1; p = 0.3801, ANCOVA; Ratio in least square means = 1.0146, 90% CI 2-sided [0.9859 to 1.0442]

2. Secondary Outcome: Maximum Skin Temperature After Rewarming (MAX)
Description: Maximum skin temperature after rewarming within 15 min after cold challenge
Time Frame: For 15 min after cold challenge (40-55 min after IMP administration)
Population: Full analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: °C
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
°C | 22.5043 (3.73) | 23.5336 (8.49)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Test type: Equivalence — Differences between treatment groups was to be detected with a power of 90% and alpha=0.1; p = 0.0356, ANCOVA; Ratio in least square means = 1.0346, 90% CI 2-sided [1.0086 to 1.0613]

3. Secondary Outcome: The Distal Dorsal Difference, Defined as the Difference in Temperature Between the Dorsum and the Finger (DDD)
Description: The distal dorsal difference, defined as the difference in temperature between the dorsum and the finger (DDD), from administration of IMP until before cold challenge (0 to 40 min)
Time Frame: Baseline, 10, 20, 30 and 40 min
Population: The full analysis set
Measure: Mean (Standard Error); unit: °C
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
°C
  Baseline | -2.810 (0.3375) | -2.4215 (0.4950)
  10 min | -3.2378 (0.3045) | -3.395 (0.4580)
  20 min | -3.0596 (0.2323) | -3.1419 (0.4792)
  30 min | -3.1005 (0.1903) | -3.0347 (0.4037)
  40 min | -2.7921 (0.1918) | -2.9448 (0.333)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Analysis at the 10 min point; Test type: Equivalence — Differences between treatment groups was to be detected with a power of 90% and alpha=0.1; p = 0.0154, ANCOVA; Difference in least square means = -0.4991, 90% CI 2-sided [-0.8234 to -0.1749]

4. Secondary Outcome: Gradient of Rewarming in the First 2 Minutes Post-cold Challenge (GRAD)
Time Frame: 2 min after cold challenge (40-42 min after IMP administration)
Population: The full analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: °C/min
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
°C/min | 0.5412 (42.26) | 0.4482 (39.35)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Test type: Equivalence — Differences between treatment groups was to be detected with a power of 90% and alpha=0.1; p = 0.282, ANCOVA; Ratio in least square means = 0.8301, 90% CI 2-sided [0.6206 to 1.1102]

5. Other Pre Specified Outcome: Change in Finger Temperature From Intake of IMP to Start of Cold Challenge
Time Frame: From intake of IMP to start of cold challenge (0-40 min)
Population: The full analysis set
Measure: Mean (Standard Error); unit: °C
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
°C | -0.697 (0.471) | -1.347 (0.343)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Test type: Equivalence — Differences between treatment groups was to be detected with a power of 90% and alpha=0.1; p = 0.3722, ANCOVA; Difference in least square means = -0.3989, 90% CI 2-sided [-1.1718 to 0.3739]

6. Other Pre Specified Outcome: Nailfold Capillaroscopy (Including Red Blood Cell Velocity Measurements)
Description: Nailfold capillaroscopy mean velocity was measured as red blood cell velocity before cold challenge and post recovery
Time Frame: Before cold challenge (at 40 min) and post-recovery (at 55 min)
Population: The full analysis set
Measure: Mean (Standard Error); unit: mm/sec
Arm/Group | Placebo | C21 200 mg
Number analyzed (Participants) | 12 | 12
mm/sec
  Baseline | 0.122 (0.042) | 0.369 (0.193)
  Before cold | 0.302 (0.175) | 0.207 (0.054)
  Post recovery | 0.318 (0.140) | 0.323 (0.149)
Statistical Analysis 1: Comparison: Placebo vs C21 200 mg; Analysis of capillaroscopy before cold; Test type: Equivalence — Differences between treatment groups was to be detected with a power of 90% and alpha=0.1; p = 0.4982, ANCOVA; Difference in least square means = -0.109, 90% CI 2-sided [-0.4074 to 0.1895]
Statistical Analysis 2: Comparison: Placebo vs C21 200 mg; Analysis of capillaroscopy post recovery; Test type: Equivalence — A difference between treatment groups was detected with a power of 90% and alpha=0.1; p = 0.6219, ANCOVA; Difference in least square means = -0.0637, 90% CI 2-sided [-0.3037 to 0.1763]

ADVERSE EVENTS:
Time Frame: From signing of informed consent through study completion, an average of 30 days
Description: At each visit the subject was asked about adverse events (AEs) in an objective manner, e.g.: "Have you experienced any problems since the last visit?"
Arm/Group | Placebo | C21 200 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | C21 200 mg (N=12)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT04388176/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04388176/SAP_001.pdf